CLINICAL TRIAL: NCT03660007
Title: Association of Pulmonary and Venous Thromboembolism in IVF Pregnancies After Fresh and Frozen Embryo Transfer: a Population-based Cohort Study
Brief Title: Incidence of Pulmonary and Venous Thromboembolism in IVF Pregnancies After Fresh and Frozen Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Henriksson, Professor, Karolinska Institutet
Other Study IDs: Fresh or Frozen IVF
Record Dates: First submitted 2018-08-30; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Assisted Reproductive Techniques; Pregnancy; Pulmonary Embolism; Venous Thromboembolism; Fresh Embryo Transfer; Frozen Embryo Transfer
Keywords: In vitro fertilization; Assisted Reproductive Techniques; Pulmonary embolism; Venous Thromboembolism; Pregnancy
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fresh embryo transfer: This exposure is an IVF pregnancy with fresh embryo transfer performed directly after ovarian stimulation
  Interventions: Procedure: Fresh or frozen embryo transfer IVF
- Frozen embryo transfer: This exposure is an IVF pregnancy with frozen embryo transfer, which was thawed and transferred in a later, non-stimulated cycle
  Interventions: Procedure: Fresh or frozen embryo transfer IVF
- Natural pregnancy: Spontaneous pregnancy without IVF

INTERVENTIONS:
Procedure: Fresh or frozen embryo transfer IVF
  Groups: Fresh embryo transfer; Frozen embryo transfer

SUMMARY:
In vitro fertilization (IVF) is associated with an increased risk of venous thromboembolism and in particular pulmonary embolism during the first trimester. It is not known whether this increased risk of pulmonary embolism is present both after fresh and frozen embryo transfer.

Objective: To assess whether the risk of pulmonary embolism and venous thromboembolism during the first trimester of IVF pregnancies is associated with both fresh and frozen embryo transfer.

A population-based cohort study with linked data from nationwide registries on women in Sweden giving birth to their first child 1992-2012

DETAILED DESCRIPTION:
A population-based cohort study with data prospectively collected in the nationwide registries in Sweden. Through the national registries the investigators collect data on all women with a child born in Sweden between 1992-2012 and these will be linked to data from the registries by the use of the unique personal identity number.

Study population All women who gave birth at the age of 15-50 years to their first child from the 1st of January 1992 until the 31st of December 2012 comprise the study population. Women will be categorized as either giving birth after IVF or natural conception pregnancies. Data on whether IVF was performed by the use of fresh or frozen embryo transfer will be retrieved.

The registries The national registries in Sweden are considered to have good coverage and validity in general and the Swedish Medical Birth Register (MBR) by the National Board of Health and Welfare in Sweden includes annually 97-99.5 % of all child births in Sweden, up until 2005 all live child births and stillborn from week 28 and thereafter including all child births from week 22. From the MBR and the Swedish national quality registry of assisted reproductive technology, the Q-IVF, the investigators collect information on pre-pregnancy and pregnancy variables. From the Patient registry (PR) ICD codes for PE and overall VTE will be retrieved and from the Swedish register of Education completed years at school and finally from the Swedish Cause of Death Register data on causes of deaths .

Time periods - pregnancy length, the trimesters and postpartum. The follow-up period is from the estimated start of pregnancy until day 42 after delivery, i.e. six weeks postpartum or until an event of PE or other VTE occurred before the end of that period. When determining the trimesters, the best estimation of pregnancy length from the MBR that estimates the days of pregnancy by primary ultrasound will be used or when this is missing by calculation of the first day of the last period. Start of pregnancy is defined as the date of delivery minus the precalculated best estimation of the pregnancy length found in the MBR. Regarding trimesters and postpartum the first trimester is defined to comprise the start of pregnancy, day 0 until day 90, the second trimester from day 91 until day 181 and the third trimester from day 182 until three days before delivery date. Delivery and postpartum period is defined to comprise two days before until six weeks after delivery date, since labor often starts 1-2 days before the actual delivery. Women with pregnancy length exceeding 300 days are to be excluded, considered as extreme values.

Exposures - IVF with fresh or frozen embryo transfer The exposures are either an IVF pregnancy with fresh embryo transfer performed directly after ovarian stimulation or an IVF pregnancy with frozen embryo transfer, which was thawed and transferred in a later, non-stimulated cycle. These exposures will be compared to a control group of non-exposed women which consists of all pregnant women not listed in the MBR or the IVF-registries and thus considered to be spontaneously conceived, here referred to as natural pregnancy.

Outcome - first incident pulmonary embolism or overall venous thromboembolism The outcome is the occurrence of the first incident PE or first incident VTE during pregnancy or postpartum. All women with pre-pregnancy events are excluded.

The diagnoses of PE and DVT will be defined in the PR with data from 1987 on national inpatient care and from 1997 also outpatient and diagnoses based on the International classification of diseases, ICD. The investigators will use the 8th edition, ICD-8 (1969-1986), for previous diagnoses and exclusions of pre-pregnancy venous thromboembolism and the ninth, ICD-9 (1987-1996), and the tenth edition, ICD-10 (1997--), for both previous and incident diagnoses.

The investigators will use all diagnosis codes for PE (ICD-8: 450.01-03, 450.09, 673.98-99; ICD-9: 415B, 673C; ICD-10: I26.0, I26.9, O882), DVT (ICD-8: 451.00, 451.98-99, 671.01-02, 671.08-09; ICD-9: 451B; ICD-10: I80.1-3, I80.8-9, O22.3, O87.1), portal vein thrombosis (ICD-8 453.09; ICD-9: 452; ICD-10: I81.9), vena cava thrombosis (ICD-8; ICD-9: 453C; ICD-10: I82.2), renal thrombosis (ICD-8; ICD-9: 453D; ICD-10: I82.3), cerebral vein thrombosis (ICD-8: 321.00, 321.09; ICD-9: 325; ICD-10: O22.5, O87.3 and diagnoses codes for other localizations of DVT or emboli (ICD-8: 453.09; ICD-9: 453W, 453X, 671F; ICD-10: I82.8-9, O87.9).

Other predictors or potential confounding factors. The investigators will adjust for potential confounding factors; age, calendar year of delivery, body mass index (BMI), multiple birth, smoking, country of birth and education level. Age is one of the strongest known risk factors for VTE. BMI of 30 or more is a known risk factor for VTE. Another risk factor for VTE is parity, which is one of the reasons why the investigators in this study choose to study only the first child birth in all women in contrast to a previous study where women were included with their first IVF pregnancy. Thus, that study also included women who had given birth to a child before without known IVF with adjustments performed in the statistical analysis for parity.

The continuous variables are to be categorized as follows, age at delivery (<25, 25-29, 30-34, ≥35 years), pre-pregnancy BMI (<25, 25-29 or ≥30 kg/m2), educational level recorded as number of school years (≤9 years -compulsory school, 10-12 years - upper secondary school, >12 years -University level), pre-pregnancy cigarette smoking status (yes/no). Country of birth is either Sweden or other country.

Statistical analyses:

Baseline characteristics of women are to be reported as frequencies and percentages for categorical variables and as median and interquartile range for continuous variables.

Cox regression models are to be used to estimate hazard ratios (HRs) and 95% confidence intervals (CI) in order to assess the association between exposure (IVF with fresh or frozen embryo transfer versus the referent group with natural conception) and each of the two study outcomes. First, HRs are to be estimated under a proportional hazard assumption for the entire pregnancy duration, including the postpartum period. Then, this assumption will be relaxed by allowing the HRs to vary over the different trimesters and the postpartum period by means of a time-dependent Cox regression model. Models are to be adjusted for potential confounders as described above.

ELIGIBILITY:
Inclusion Criteria:

* Women who had given birth to a first child

Exclusion Criteria:

* Women with previous pregnancies

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All Swedish women who had given birth at the age of 15-50 years to a first child from the 1st of January 1992 until the 31st of December 2012 .
Sampling Method: Non-Probability Sample
Enrollment: 902891 (Actual)
Dates: Start 1992-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
First incident pulmonary embolism | Estimated start of pregnancy until day 90
  Pulmonary embolism during the period from start of pregnancy until pregnancy day 90

SECONDARY OUTCOMES:
First incident venous thromboembolism | Estimated start of pregnancy until day 90
  Venous thromboembolism during the period from start of pregnancy until pregnancy day 90

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olausson N, Discacciati A, Nyman AI, Lundberg F, Hovatta O, Westerlund E, Wallen HN, Mobarrez F, Bottai M, Ekbom A, Henriksson P. Incidence of pulmonary and venous thromboembolism in pregnancies after in vitro fertilization with fresh respectively frozen-thawed embryo transfer: Nationwide cohort study. J Thromb Haemost. 2020 Aug;18(8):1965-1973. doi: 10.1111/jth.14840. Epub 2020 May 11. PMID 32289205